CLINICAL TRIAL: NCT06539078
Title: Exercise as a Countermeasure Against the Effects of Ageing on Muscle Mitochondria, Diffusive Oxygen Transport and Muscle Volume
Brief Title: Skeletal Muscle Mitochondria in Ageing
Acronym: AGAMEMNON
Status: Recruiting | Type: Observational
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Dr Richie Goulding, Principal Investigator, VU University of Amsterdam
Other Study IDs: 2023.0746
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Aging
Keywords: Exercise; Mitochondria; Skeletal muscle
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test; Dental Occlusion; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Muscle biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young, sedentary participants: * Aged between 18-30 years
  * Male or female
  * Not currently engaging in any formal exercise training or competitive sports
  * No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise
  Interventions: Other: Maximal exercise test; Other: 3D Ultrasound; Other: Dynamometry; Other: Exercise test and occlusions; Other: Exercise test in MRI; Procedure: Muscle biopsy
- Young endurance-trained participants: * Aged between 18-30 years
  * Male or female
  * Currently engaging in formal training (at least 3 times per week) in competitive endurance sports (i.e. running, cycling, swimming, triathlon, etc.)
  * No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise
  Interventions: Other: Maximal exercise test; Other: 3D Ultrasound; Other: Dynamometry; Other: Exercise test and occlusions; Other: Exercise test in MRI; Procedure: Muscle biopsy
- Middle-aged, sedentary participants: * Aged between 50-65 years
  * Male or female
  * Not currently engaging in any formal exercise training or competitive sports
  * No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise
  Interventions: Other: Maximal exercise test; Other: 3D Ultrasound; Other: Dynamometry; Other: Exercise test and occlusions; Other: Exercise test in MRI; Procedure: Muscle biopsy
- Middle-aged endurance-trained participants: * Aged between 50-65 years
  * Male or female
  * Currently engaging in formal training (at least 3 times per week) in competitive endurance sports (i.e. running, cycling, swimming, triathlon, etc.)
  * No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise
  Interventions: Other: Maximal exercise test; Other: 3D Ultrasound; Other: Dynamometry; Other: Exercise test and occlusions; Other: Exercise test in MRI; Procedure: Muscle biopsy

INTERVENTIONS:
Other: Maximal exercise test — Participants will undertake an incremental ramp test on a cycle ergometer to determine maximal oxygen uptake (V̇O2max) and the gas exchange threshold (GET). Throughout the exercise test, muscle oxygenation and deoxygenation will be monitored by NIRS.
Other: 3D Ultrasound — Muscle volume and morphological characteristics will be assessed via 3D ultrasound imaging.
Other: Dynamometry — To determine the contractile properties of the knee extensors, participants will perform maximal isometric and isoinertial contractions of the knee extensors on a dynamometer.
Other: Exercise test and occlusions — Participants will perform a series of moderate-intensity constant power output exercise bouts on a cycle ergometer following which the recovery rates of muscle V̇O2 will be determined via a series of intermittent arterial occlusions. Throughout all tests, pulmonary gas exchange and ventilation will be determined and muscle oxygenation and deoxygenation will be monitored by NIRS.
Other: Exercise test in MRI — Exercise will be performed on a custom-built magnetic resonance-compatible cycle ergometer in supine position for determination of muscle phosphocreatine recovery kinetics using 31phosphorous magnetic resonance spectroscopy [31P-MRS].
Procedure: Muscle biopsy — A muscle biopsy will be obtained from the vastus lateralis using a modified Bergström needle technique with suction.

SUMMARY:
Healthy ageing is associated with the loss of muscle mass and physical function. As a result, older people are limited in their independence. The aging of muscles typically begins around the age of 30. From this age onward, muscle strength, muscle mass, and the maximum oxygen uptake of muscles decrease. The reasons for this are not entirely clear, but it seems to be partly related to how oxygen moves from our blood vessels to the muscles and how muscles burn energy. The precise role of age and physical fitness, as well as whether exercise can counteract the effects of ageing, is still unknown. Therefore, in this study, we aim to investigate the muscle function of both physically active and inactive young and middle-aged individuals. We hypothesise that endurance training can mitigate some of the effects of ageing.

DETAILED DESCRIPTION:
Healthy ageing is associated with a loss of muscle mass and physical function. This loss of physical function is underpinned by reductions in characteristics such as muscle strength, power, and maximal oxygen uptake (V̇O2max; reflecting exercise capacity). However, the causal contributors to these age-associated impairments, and the role of exercise training status in mitigating them, remain poorly defined. Skeletal muscle mitochondrial function has been proposed to be a key contributor to age-associated effects on physical function, however many conflicting results are present in the extant human literature. Moreover, diffusion of oxygen from capillaries to mitochondria is a key determinant of V̇O2max, however, whether the skeletal muscle diffusive capacity for oxygen (DmO2) declines with age is unknown. A new technique utilizing near-infrared spectroscopy (NIRS) will enable the non-invasive assessment of skeletal muscle diffusive capacity in young and elderly subjects for the first time to resolve this issue. The primary aims of this study are therefore to 1) compare DmO2 derived via NIRS between young sedentary, young endurance-trained, older sedentary, and older endurance-trained subjects; 2) to compare non-invasive (i.e. with NIRS and 31phosphorous magnetic resonance spectroscopy [31P-MRS]) and invasive (i.e. measures of mitochondrial morphology and respiration obtained by skeletal muscle biopsy) markers of mitochondrial function between the same groups, and 3) to assess the relationships between DmO2, mitochondrial measures and assessments of capillarization with functional measurements of muscle strength, power, and V̇O2max.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, young sedentary participants must meet all of the following criteria:

* Aged between 18-30 years
* Male or female
* Not currently engaging in any formal exercise training or competitive sports
* No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise

In order to be eligible to participate in this study, young trained participants must meet all of the following criteria:

* Aged between 18-30 years
* Male or female
* Currently engaging in formal training (at least 3 times per week) in competitive endurance sports
* No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise

In order to be eligible to participate in this study, older sedentary participants must meet all of the following criteria:

* Aged between 50-65 years
* Male or female
* Not currently engaging in any formal exercise training or competitive sports
* No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise

In order to be eligible to participate in this study, older trained participants must meet all of the following criteria:

* Aged between 50-65 years
* Male or female
* Currently engaging in formal training (at least 3 times per week) in competitive endurance sports
* No chronic health conditions likely to affect exercise tolerance or the physiological responses to exercise

Exclusion Criteria:

* Age that falls outside of 18-30 years (young groups) or 50-65 years (middle-aged groups)
* Inability to provide informed consent
* History of claustrophobia
* Ineligibility to perform the exercise test described in this study protocol or follow instructions
* Taking any medications known to interfere with the physiological responses to exercise, e.g. e.g. systemic corticosteroids, statins, SGLT2 inhibitors, GLP1 receptor agonists
* Contraindication for MRI (e.g. pacemaker, claustrophobia)
* Being under investigation for non-diagnosed disease at the time of investigation
* Body Mass Index (BMI) >30 due to adiposity, since this is known to cause difficulties in obtaining muscle biopsies and NIRS measurements
* Pregnancy
* Are current smokers or have been a regular smoker within the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 sedentary and 15 endurance-trained young and middle-aged individuals will be recruited per age group (i.e. a total of 60 individuals spanning 4 groups). An equal balance of the sexes will be aimed for in each group. All participants will be recruited from specific social media groups, through personal networks of friends, family and colleagues, flyers and posters at local sports clubs and on the VU Campus. All testing will be conducted at the VU or in the Department of Radiology and Nuclear Medicine at Amsterdam UMC location AMC. Therefore, participants should be currently residing in or willing to travel to Amsterdam.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (V̇O2max) | Baseline (visit 1)
  ml/min/kg
Muscle volume | Baseline (visit 1)
  cm^3
Muscle strength | Baseline (visit 1)
  Newton-metre (Nm)
Muscle power | Baseline (visit 1)
  Watt (W)
Muscle diffusing capacity for oxygen (DmO2) | Baseline (visit 1) and visit 2-4. In total 4 weeks.
  Differences in recovery constant k (min-1) obtained under conditions of high, medium or low O2 availability
Muscle mitochondrial fragmentation index (A.U.) | Visit 6 muscle biopsy (+/- after 4 weeks).
  Degree of fragmentation of the mitochondrial pool.

SECONDARY OUTCOMES:
Gas exchange and ventilatory variables (gas exchange threshold, respiratory compensation point, maximal ventilation) | Baseline (visit 1)
  L/min
(Peak) power output | Baseline (visit 1)
  Watt (W)
Mean response time of the V̇O2 slope during ramp exercise | Baseline (visit 1)
  sec
(Maximum) heart rate (HR) | Baseline (visit 1) and during visit 2-4 (max 4 weeks in total)
  beats per minute (bpm)
Maximal O2 pulse | Baseline (visit 1)
  ml/beat
Slope of ventilation (VE) versus carbon dioxide (VCO2) output during ramp exercise (i.e. ventilatory efficiency) | Baseline (visit 1)
  V̇E/V̇CO2 slope
V̇O2/HR slope during ramp exercise | Baseline (visit 1)
  beats/L/min
Maximal respiratory exchange ratio (RER) | Baseline (visit 1)
  RER = VCO2/VO2
Maximal ventilatory equivalents | Baseline (visit 1)
  VE/VCO2 and VE/VO2
Maximal end-tidal pressures for oxygen (O2) and carbon dioxide (CO2) | Baseline (visit 1)
  mmHg
Capillary lactate concentration | Baseline (visit 1)
  mmol/L
Maximal respiratory frequency | Baseline (visit 1)
  breaths/min
Pulmonary oxygen uptake - baseline and steady state V̇O2 | Baseline (visit 1) and visit 2-4 (max 4 weeks in total)
  L/min
Pulmonary oxygen uptake kinetics - Phase II V̇O2 time constant and time delay | Visit 2-4 (max 4 weeks in total)
  sec
Pulmonary oxygen uptake kinetics - Phase II V̇O2 amplitude | Visit 2-4 (max 4 weeks in total)
  L/min
Concentrations of NIRS derived muscle oxy- and deoxygenated [haemoglobin + myoglobin] (HbO2, Hbb) and tissue saturation index (TSI). | Baseline (visit 1) and visit 2-4 (max 4 weeks in total)
  HbO2 and Hbb: % maximal value, TSI (%) = HbO2/(HbO2+Hbb) For all variables resting concentration, baseline cycling concentration, (sub)maximal exercise concentration will be reported.
NIRS derived muscle oxy- and deoxygenated [haemoglobin + myoglobin] (HbO2, Hbb) and tissue saturation index (TSI) versus relative and absolute work rate. | Baseline (visit 1)
  HbO2 and Hbb: % maximal value, TSI (%) = HbO2/(HbO2+Hbb) versus relative (%max) and absolute power output (W) Relative and absolute work rates comparisons will be reported for all variables: resting concentration, baseline cycling concentration, (sub)maximal exercise concentration.
Initial and secondary slope of increase during incremental exercise will be reported for NIRS derived muscle oxy- and deoxygenated [haemoglobin + myoglobin] (HbO2, Hbb) and tissue saturation index (TSI) versus relative work rate. | Baseline (visit 1)
  concentration[Hbb/HbO2/TSI]%/delta%peak power(W)
Initial and secondary slope during incremental exercise will be reported for NIRS derived muscle oxy- and deoxygenated [haemoglobin + myoglobin] (HbO2, Hbb) and tissue saturation index (TSI) versus absolute work rate. | Baseline (visit 1)
  concentration[Hbb/HbO2/TSI]%/deltaW
Muscle (de)oxygenation breakpoint during incremental exercise | Baseline (visit 1)
  Power output (W) and maximal oxygen uptake (L/min)
Rate constant of mV̇O2 recovery kinetics under conditions of high, medium and low O2 availability | Baseline (visit 1)
  sec
Muscle morphology - Fascicle length | Baseline (visit 1)
  cm
Muscle morphology - pennation angle | Baseline (visit 1)
  degrees
Muscle morphology - (effective) physiological cross-sectional area (PCSA) | Baseline (visit 1)
  cm2
Muscle morphology - vastus lateralis specific force | Baseline (visit 1)
  N/cm2
Muscle morphology - estimated muscle fiber number | Baseline (visit 1)
  PCSA/muscle fiber cross-sectional area
Adipose tissue thickness at the site of NIRS measurement | Baseline (visit 1)
  mm
Mitochondrial respiratory function (background, LEAK, N-linked respiration, OXPHOS, ETS, succinate (S) + rotenone (ROT)-linked uncoupled respiration, ) | Visit 6 muscle biopsy (+/- after 4 weeks).
  pmol/s/mg
Respiratory control ratios | Visit 6 muscle biopsy (+/- after 4 weeks).
  OXPHOS/ETS, LEAK/ETS, LEAK/OXPHOS, LEAK/NADH-linked, ROT+S/ETS, (OXPHOS-LEAK)/ETS, (OXPHOS-LEAK)/OXPHOS, (ETS-LEAK)/ETS, (ETS-OXPHOS)/ETS
Intrinsic mitochondrial respiration (each respiratory state outlined below will be normalised to mitochondrial volume density) | Visit 6 muscle biopsy (+/- after 4 weeks).
  (pmol/s/mg)/mitochondrial area density (%) For: background, LEAK, N-linked respiration, OXPHOS, ETS, succinate + rotenone-linked uncoupled respiration
31P-MRS-derived mitochondrial bioenergetic function - resting and steady-state exercising concentrations and amplitude of exercise-induced changes of skeletal muscle Phosphocreatine [PCr], [inorganic phosphate] and pH | Visit 5 MRI
  mM pH = unitless
31P-MRS-derived mitochondrial bioenergetic function rate constant of PCr | Visit 5 MRI
  Rate constant of Phosphocreatine [PCr] on- and off-kinetics (sec)
31P-MRS-derived mitochondrial bioenergetic function - maximal rate of oxidative ATP synthesis | Visit 5 MRI
  mM/s
Muscle fiber type distribution | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  Type I, IIa, IIx and hybrid fiber-type proportions (%)
(mean) fiber cross-sectional area, also fiber type specific | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  um
Weighted fiber cross-sectional area | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  um2
Mean and fiber type specific succinate dehydrogenase activity | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  A660/um/s
Integrated fiber succinate dehydrogenase activity | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  A660.um/s
Mean and fiber type specific myoglobin concentrations | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  mM
Muscle capillarization - capillary density | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  number of capillaries/mm2
Muscle capillarization - capillary-to-fiber ratio | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  capillary-to-fiber ratio
Muscle capillarization - mean number of capillaries surrounding a fiber (CAF) | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  number of capillaries
Muscle capillarization - mean number of capillaries surrounding a fiber in relation to fiber area (CAFA) | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  number of capillaries/um2
Muscle capillarization - capillary-to fiber-perimeter exchange index (CFPE) | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  CFPE (unitless)
Muscle capillarization - length of capillaries relative to fiber perimeter (LC/PF) | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  percentage (%)
Muscle capillarization - sarcomere length | Visit 6 muscle biopsy (+/- after 4 weeks) - staining within time window of 2 years.
  um
Mitochondrial dynamics proteins (Mfn1, Mfn2, OPA1, Drp1, Parkin, PINK1, Fis1, MTFP1, NRF1&2, PGC1a, TFAM, OXPHOS protein content (complexes I-V and total protein content) | Visit 6 muscle biopsy (+/- after 4 weeks) - western blot within time window of 2 years.
  ug/mg loaded sample
Physical activity status - pedometer | Baseline 7 days
  Number of steps per day
Mitochondrial area density | Visit 6 muscle biopsy (+/- after 4 weeks) - electron microscopy (EM) within time window of 2 years.
  Percentage (%)
Mitochondrial volume density | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  um3.um3.10^2
Mitochondrial number | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  number/um2
Mitochondrial area | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  um2
Mitochondrial height, width, perimeter and maximal+minimal Feret's diameter | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  um
Mitochondrial surface area-to-volume ratio | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  um/um^2
Mitochondrial circularity | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  Circularity (AU)
Mitochondrial roundness | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  Roundness (AU)
Mitochondrial aspect ratio | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  Aspect ratio (AU)
Mitochondrial cristae area density | Visit 6 muscle biopsy (+/- after 4 weeks) - EM within time window of 2 years.
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Richie Goulding, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No